CLINICAL TRIAL: NCT02045173
Title: Screening for Sleep-disordered Breathing in Routine Cardiology Practice: Validation of the Apnea + Hypopnea Detection by an Implantable Cardioverter Defibrillator (ICD) or Cardiac Resynchronization Therapy-defibrillator (CRT-D) With Impedance-based Respiration Sensor (ApneaScanTM)
Brief Title: Automate Detection of Sleep Apnea by ApneascanTM
Acronym: AIRLESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1332
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Sleep Apnea; Arrhythmias
Keywords: Sleep apnea, Arrhythmias, Heart Failure, ICD, CRT-D, Apneascan
MeSH Terms: conditions — Sleep Apnea Syndromes; Arrhythmias, Cardiac; Heart Failure | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apneascan TM (Other): autoscoring algorithms of the Apneascan TM compared to the polysomnography or polygraphy
  Interventions: Other: Apneascan TM; Device: Polysomnography/polygraphy

INTERVENTIONS:
Other: Apneascan TM — Autoscoring algorithms with automatical detection of sleep apnea by the Apneascan TM
Device: Polysomnography/polygraphy — 1 night polysomnography/polygraphy

SUMMARY:
The purpose of the study is to compare, three months after implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy-defibrillator (CRT-D), the apnea-hypopnea index (AHI) obtained from conventional in-lab NPSG/NPG (AHIPSG) with similar indices obtained from autoscoring algorithms of the ApneaScan™, an implantable impedance-based respiration sensor (AHIAS).

DETAILED DESCRIPTION:
This is a prospective, multi center, phase-IV with blinded analysis and central reading of polysomnography trial.

The study is performed in patients with a standard CRT-D or Implantable Cardioverter Defibrillator (ICD) devices indication. A total of 160 subjects will be recruited in France. The study duration is 03 months for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged > 18 years old
* Current ICD or CRT-D device-based guidelines indication (for primo-implantation)
* patients with optimal recommended medical therapy
* Patient willing and able of undergoing the device implant procedure
* Patient willing and able of undergoing the LATITUDE® NXT Patient Management system procedure
* Patient willing and able to complete the requirements of the study including the signature of the Informed Consent after full explanation of the study by the investigator prior to participation.

Exclusion Criteria:

* Obstructive lung disease as defined by a FEV1/FVC less than 70%
* Obesity hypoventilation syndrome
* Treated sleep disorders breathing
* Cardiac surgery scheduled or strong likelihood of cardiac surgery 4 months after enrollment
* Life expectancy less than 1 year
* Inability to complete overnight PSG as defined by the protocol
* Patient who are or suspected to be pregnant and or plan to become pregnant
* Patient protected by the Law, under guardianship or curators
* Concomitant participation in an interventional biomedical research trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index obtained from polysomnography or polygraphy and from autoscoring algorithms of the ApneaScan™ implantable impedance respiration sensor | Prior the ICD or CRT-D implantation and up to 3 months

SECONDARY OUTCOMES:
Malignant arrhythmogenic events detected daily by the ICD / CRT-D (AF, ES, supraventricular tachycardia, sustained and non sustained ventricular tachycardia, VF) and night by night AHI assessed by the ApneascanTM | baseline and up to 3 months
Weekly weight readings automatically and wirelessly sent to the LATITUDE(C) | Baseline and Up to 3 months
Apnea and Hypopnea index measured 3 months after ICR or CRT-D implantation compared to the Apnea and Hypopnea index measured at baseline by the polysomnography or polygraphy | Prior the ICD or CRT-D implantation and up to 3 months

OTHER OUTCOMES:
Evolution night by night of AHI obtained from autoscoring algorithms of the ApneaScan™ implantable impedance respiration sensor | From ICD or CRT-D implantation and up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis PEPIN, MD, PhD, Principal Investigator — Grenoble Hospital University; Pascal DEFAYE, MD, Principal Investigator — Grenoble Hospital University
Locations (5):
- France (5):
  - CHU de Grenoble, Grenoble
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hopital Barbois, Nancy
  - Clinique Pasteur, Toulouse
  - Hôpital Trousseau, Tours